CLINICAL TRIAL: NCT02383823
Title: Postprandial Lipidemia and Glucose Metabolism After a Meal With Different Types of Fat, Estrogen Treatment, Age and Gender in Healthy Subjects
Brief Title: Postprandial Lipidemia After a Meal With Different Types of Fat, Estrogen Treatment, Age and Gender in Healthy Subjects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never started the inclusion
Sponsor: Herning Hospital (Other)
Collaborators: Sygehus Lillebaelt (Other)
Responsible Party: Principal Investigator, Finn Lauszus, Associate Professor, Research Specialist, Senoir Consultant, Herning Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: M-2104-99
Record Dates: First submitted 2015-02-16; First posted 2015-03-09 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Menopause
Keywords: glucose, cholesterol, estrogen, gender, age
MeSH Terms: conditions — Coitus | interventions — Estrogens; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Estrogens in menopausal women (Active Comparator): Crossover of estrogens or placebo in random order, either 2 mg estradiol or placebo in three months in random sequence, age span 45-55
  Interventions: Drug: Estrogens
- Menopausal men (No Intervention): comparative to menopausal women, age span 45-55
- Elderly women (No Intervention): comparative to menopausal women, age span 65-80
- Elderly men (No Intervention): comparative to menopausal women, age span 65-80
- Placebo in menopausal women (Placebo Comparator): Crossover of estrogen or placebo in random order, either 2 mg estrogen or placebo in three months in random sequence, age span 45-55
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Estrogens — Crossover study of estrogen or placebo in random order in menopausal women
  Other Names: Estradiol
  Arms: Estrogens in menopausal women
Other: Placebo — Crossover study of placebo or estrogen in random order in menopausal women
  Arms: Placebo in menopausal women

SUMMARY:
The study examines the effect of hormone replacement in postmenopausal women compared to men, 55 years of age, and in the elderly without hormone replacement of both sexes. The lipid and glucose metabolism is evaluated during treatment and placebo with a meal with mashed potatoes and different types of fat. Glucose, insulin, triglyceride, total cholesterol, LDL and HDL cholesterol, free fatty acids and coagulation parameters are measured.

During menopause the women reduce their levels of estrogen and their risk of cardiovascular disease rises to the men's level. This effect on mortality and morbidity can probably be reduced by hormone therapy.

DETAILED DESCRIPTION:
The experiment illustrates the gender, age and estrogen influence the acute metabolic responses after meal consisting of mashed potatoes added different types of fat. The reason is that the distribution of macronutrients are often not equal to the ideal and fat intake in Western countries is well above the recommended maximum of 30%. A high fat intake -especially saturated fat -increases the risk of ischemic heart disease significantly and HDL cholesterol levels are determined by the postprandial lipid response. The negative correlation between HDL cholesterol and ischemic heart disease can apparently be attributed to a strong positive correlation between postprandial lipidemia and ischemic heart disease.

Diet has an important role in both the development and treatment of diseases such as type 2 diabetes, elevated blood cholesterol, and obesity. It is recommended today to eat a high-carbohydrate and low-fat diet with reduced energy in these patients. Postprandial lipid in the blood after fat meals expected to be gender-specific, since men's total and LDL-cholesterol and triglycerides are higher than in women of childbearing age. Menopause reduces women's estrogen levels and increase their risk of cardiovascular disease to men's level. This effect on morbidity and mortality is influenced probably by hormone replacement. What influence it has on the postprandial responses is uncertain. The haemostatic system plays an important role in the development of ischemic heart disease and in acute conditions such as acute myocardial infarction, unstable angina, and sudden cardiac death. Fat-rich meals induces an acute activation of coagulation factors and postprandial lipid levels in the blood are essential to the development of atherosclerosis and coagulation activation 4 to 8 hours after a meal. The influence of gender, age, estrogen and different fat types of these conditions are not yet fully elucidated. The investigators believe it is important to investigate the effect of addition of different types of fat to a starchy meal on blood glucose, insulin and lipid levels in healthy subjects, since the metabolic responses today considered closely associated to the development of atherosclerosis and type 2 diabetes.

The investigators therefore wish to investigate the effect of hormones in postmenopausal women compared to men and to assess the effect of age in both sexes of acute metabolic responses by examining the age groups 45-55 (40 women in total in 5 different hormone treatments and 8 men) and 65-80 years (16 in total, 8 of each gender).

The effect is assessed on glycemic response, insulin, triglyceride, total cholesterol, LDL and HDL cholesterol, apo-lipoprotein, free fatty acids and coagulation parameters (von Willebrand factor, Factor VII, Factor VIIa, Plasminogen activator inhibitor-1, fibrinogen, tissue thromboplastin, fibrin).

ELIGIBILITY:
Inclusion Criteria:

* Men, age 45-55
* Men age 65-80
* Women age 45-55: The menopausal women's follicle stimulating hormone and luteinizing hormone levels should be above 40 nmol/l
* Women age 65-80

Exclusion Criteria:

* hypercholesterolemia,
* hypertension,
* substance abuse or alcohol abuse
* recognized renal, hepatic, cardiac and metabolic disorders,
* thromboembolic diseases,
* active cancer of the uterus or breast or
* other hormone replacement therapy.
* If pronounced side effects of hormone treatment, the subject is omitted from the trial

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Postprandial lipidemia | Three months of estrogen treatment
  Comparison of area under curve of lipids after estrogen treatment with no treatment, gender, and age: Cholesterol, LDL; HDL, TG; FFA: Unit: mmol/L*480 min

SECONDARY OUTCOMES:
Postprandial glucose and insulin | Three months of estrogen treatment
  Comparison of area under curve of glucose (mmol/L * 480 min) and insulin (micro-equivalents/L* 480 min) after estrogen treatment with no treatment, gender, and age

CONTACTS AND LOCATIONS:
Overall Officials: Finn F Lauszus, MD,PhD, Principal Investigator — Herning Hospital, Denmark
Locations (1):
- Gynecology Dept. Herning Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No